CLINICAL TRIAL: NCT03384654
Title: An Open-label, Multicenter, Phase 2 Study Evaluating the Efficacy and Safety of Daratumumab in Pediatric and Young Adult Subjects >=1 and <=30 Years of Age With Relapsed/Refractory Precursor B-cell or T-cell Acute Lymphoblastic Leukemia or Lymphoblastic Lymphoma
Brief Title: A Study to Evaluate the Efficacy and Safety of Daratumumab in Pediatric and Young Adult Participants Greater Than or Equal to (>=)1 and Less Than or Equal to (<=) 30 Years of Age With Relapsed/Refractory Precursor B-cell or T-cell Acute Lymphoblastic Leukemia or Lymphoblastic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108432; 2017-003377-34 (EudraCT Number); 54767414ALL2005 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-12-20; First posted 2017-12-27 (Actual); Results first posted 2023-10-13 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Precursor Cell Lymphoblastic Leukemia-Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — daratumumab; Vincristine; Prednisone; Doxorubicin; pegaspargase; Cyclophosphamide; Cytarabine; Mercaptopurine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: B-Cell Acute Lymphoblastic Leukemia (ALL)/LL (Experimental): Cohort 1 will include participants with B cell ALL/LL in second or greater relapse or refractory to at least 2 prior induction regimens. Participant will receive daratumumab in combination with vincristine and prednisone.
  Interventions: Drug: Daratumumab; Drug: Vincristine; Drug: Prednisone
- Cohort 2: T-Cell ALL/LL (Experimental): Cohort 2 will include participants with T-cell ALL/LL in first relapse or refractory to at least 1 prior induction/consolidation regimen. Participant will receive daratumumab in combination with vincristine, prednisone, doxorubicin and peg-asparaginase in Cycle 1 and daratumumab in combination with cyclophosphamide, cytarabine, 6- mercaptopurine and methotrexate in Cycle 2.
  Interventions: Drug: Daratumumab; Drug: Vincristine; Drug: Prednisone; Drug: Doxorubicin; Biological: Peg-asparaginase; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: 6-mercaptopurine; Drug: Methotrexate

INTERVENTIONS:
Drug: Daratumumab — Participant will receive daratumumab 16 milligram per kilogram (mg/kg) in cohort 1 and cohort 2.
Drug: Vincristine — Participant will receive vincristine 1.5 milligram per meter square (mg/m^2) in cohort 1 and cohort 2.
Drug: Prednisone — Participant will receive prednisone 40 mg/m^2 in cohort 1 and cohort 2.
Drug: Doxorubicin — Participant will receive doxorubicin 60 mg/m^2 in cohort 2.
  Arms: Cohort 2: T-Cell ALL/LL
Biological: Peg-asparaginase — Participant will receive peg-asparaginase 2500 units per meter square (U/m^2) in cohort 2.
  Arms: Cohort 2: T-Cell ALL/LL
Drug: Cyclophosphamide — Participant will receive cyclophosphamide 1 gram per meter square (g/m^2) once in cohort 2.
  Arms: Cohort 2: T-Cell ALL/LL
Drug: Cytarabine — Participant will receive cytarabine 75 mg/m^2 in cohort 2.
  Arms: Cohort 2: T-Cell ALL/LL
Drug: 6-mercaptopurine — Participant will receive 6-mercaptopurine 60 mg/m^2 orally daily in cohort 2.
  Arms: Cohort 2: T-Cell ALL/LL
Drug: Methotrexate — Participant will receive methotrexate 5 g/m^2 intravenously (IV) in cohort 2.
  Arms: Cohort 2: T-Cell ALL/LL

SUMMARY:
The purpose of this study is to evaluate the efficacy of daratumumab in addition to standard chemotherapy in pediatric participants with relapsed/refractory B-cell acute lymphoblastic leukemia (ALL)/lymphoblastic lymphoma (LL) and T-cell ALL/LL as measured by the complete response (CR) rate.

DETAILED DESCRIPTION:
Screening for eligible participants will be performed within 21 days before administration of the study drug. Participants with B-cell ALL/LL will receive treatment until disease progression, unacceptable toxicity or achievement of CR followed by hematopoietic stem cell transplant (HSCT). Participants with T cell ALL/LL will receive treatment for up to 2 cycles. If disease progression is confirmed, then the participant will discontinue study treatment, complete the End of Treatment Visit, and enter the Posttreatment Period. For those participants who discontinue study drug prior to disease progression, disease evaluations will continue to be performed every 8 weeks until subsequent anticancer therapy is initiated.

ELIGIBILITY:
Inclusion Criteria:

* Documented acute lymphoblastic leukemia (ALL) or lymphoblastic lymphoma (LL) as defined by the criteria below:

  1. B-cell cohort: Stage 1; ALL in second or greater relapse or refractory to 2 prior induction regimens with greater than or equal to (>=) 5 percent (%) blasts in the bone marrow and aged 1 to less than (<) 18 years. Stage 2; ALL in second or greater relapse or refractory to 2 prior induction regimens with (>=) 5% blasts in the bone marrow and aged 1 to 30 years. LL in second or greater relapse or refractory to 2 prior induction regimens and biopsy proven and with evidence of measurable disease by radiologic criteria and aged 1 to 30 years.
  2. T-cell cohort: Stage 1; ALL in first relapse or refractory to 1 prior induction/consolidation regimen with (>=) 5% blasts in the bone marrow and aged 1 to <18 years. Stage 2; ALL in first relapse or refractory to 1 prior induction/consolidation regimen with (>=) 5% blasts in the bone marrow and aged 1 to 30 years. LL in first relapse or refractory to 1 prior induction/consolidation regimen biopsy proven and with evidence of measurable disease by radiologic criteria and aged 1 to 30 years
* Performance status greater than or equal to (>=) 70 by Lansky scale (for participants less than [<] 16 years of age) or Karnofsky scale (for participants [>=] 16 years of age)
* Adequate hematology laboratory values at Cycle 1 Day 1 pre-dosing defined as follows:

  1. Hemoglobin (>=) 7.5 gram per deciliter (g/dL) ([>=] 5 millimole per liter [mmol/L]; prior red blood cell [RBC] transfusion is permitted)
  2. Platelet count (>=) 10*10^9 per liter (L) (prior platelet transfusion is permitted)
* Adequate renal function defined as normal serum creatinine for the participant's age or creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 milliliter per minute per 1.73 square meter (mL/min/1.73 m^2) prior to enrollment
* Adequate liver function prior to enrollment defined as:

  1. Alanine aminotransferase level less than or equal to (<=) 2.5* the upper limit of normal (ULN),
  2. Aspartate aminotransferase level (<=) 2.5* ULN, and
  3. Total bilirubin (<=) 2* ULN or direct bilirubin level (<=) 2.0* ULN

Exclusion Criteria:

* Received an allogeneic hematopoietic transplant within 3 months of screening
* Active acute graft-versus-host disease of any grade or chronic graft-versus-host disease of Grade 2 or higher
* Received immunosuppression post hematopoietic transplant within 1 month of study entry
* Philadelphia chromosome positive (Ph+) B-cell ALL eligible for tyrosine kinase inhibitor therapy
* Has either of the following:

  1. Evidence of dyspnea at rest or oxygen saturation (<=) 94 percent (%).
  2. Known moderate or severe persistent asthma within the past 2 years, or uncontrolled asthma of any classification
* Received an investigational drug, was vaccinated with live attenuated vaccines, or used an invasive investigational medical device within 4 weeks before the planned first dose of study drug, or is currently being treated in an investigational study
* Known to be seropositive for human immunodeficiency virus (HIV)
* Any one of the following:

  1. Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Participants with resolved infection (ie, participants who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) levels. Those who are PCR positive will be excluded
  2. Known to be seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy)

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (53):
- United States (26):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Children's Hospital Orange County, Orange, California
  - Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children'S Healthcare Of Atlanta/Emory Univ. Dept. Of Pediatrics, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Washington Univeristy School of Medicine/ Pediatrics, St Louis, Missouri
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - New York University Langone Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Dell Children's Medical Center of Central Texas/Children's Blood and Cancer Center, Austin, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Utah Primary Children's Medical Center, Salt Lake City, Utah
  - Medical College Of Wisconsin, Milwaukee, Wisconsin
- Universitair Ziekenhuis Gent - UZ GENT, Ghent, Belgium
- France (5):
  - CHU de Bordeaux, Hopital des Enfants, Bordeaux
  - IHOPE - Hospices civils de Lyon, Lyon
  - Hopital trousseau- APHP, Paris
  - Hôpital Robert Debré, Paris
  - Hôpital D'Enfants, Vandœuvre-lès-Nancy
- Germany (3):
  - Charite-Universitätsmedizin Berlin - Berlin, Berlin
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum Munster, Münster
- Schneider Children's Medical Center, Petach Tiquva, Israel
- Italy (4):
  - Istituto Giannina Gaslini, Genova
  - Fondazione MBBM, ASST Monza, Monza
  - Ospedale Pediatrico Bambin Gesù, Roma
  - AOU Città della Salute e della Scienza di Torino, Presidio Ospedale Infantile Regina Margherita, Torino
- Princess Maxima Center, Utrecht, Netherlands
- Spain (4):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Sant Joan de Deu, Esplugues de Llobregat
  - Hosp. Infantil Univ. Nino Jesus, Madrid
  - Hosp. Univ. I Politecni La Fe, Valencia
- Karolinska University Hospital, Stockholm, Sweden
- United Kingdom (7):
  - Bristol Royal Hospital for Children, Bristol
  - Royal Hospital for Sick Children, Glasgow
  - Leeds Children's Hospital, Leeds
  - University College London Hospitals, London
  - Great Ormond Street Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - Royal Marsden Hospital, Surrey

REFERENCES:
- [Derived] Bhatla T, Hogan LE, Teachey DT, Bautista F, Moppett J, Velasco Puyo P, Micalizzi C, Rossig C, Shukla N, Gilad G, Locatelli F, Baruchel A, Zwaan CM, Bezler NS, Rubio-San-Simon A, Taussig DC, Raetz EA, Mao ZJ, Wood BL, Alvarez Arias D, Krevvata M, Nnane I, Bandyopadhyay N, Lopez Solano L, Dennis RM, Carson R, Vora A. Daratumumab in pediatric relapsed/refractory acute lymphoblastic leukemia or lymphoblastic lymphoma: the DELPHINUS study. Blood. 2024 Nov 21;144(21):2237-2247. doi: 10.1182/blood.2024024493. PMID 39158071
- [Derived] Ruhayel SD, Valvi S. Daratumumab in T-cell acute lymphoblastic leukaemia: A case report and review of the literature. Pediatr Blood Cancer. 2021 May;68(5):e28829. doi: 10.1002/pbc.28829. Epub 2020 Nov 27. No abstract available. PMID 33245179

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After enrollment of 47 participants, one participant in Cohort 1: B-cell acute lymphoblastic leukemia (ALL) (1-17 Years) was withdrawn prior to receiving treatment, and thus only 46 participants were treated in the study.
Groups:
- Cohort 1: B-cell ALL (1-17 Years): Participants with relapsed/refractory B-cell ALL received intrathecal methotrexate (MTX) 8 milligrams (mg): 1 to less than (<) 2 years, 10 mg: 2 to <3 years, 12 mg: 3 to <9 years and 15 mg: greater than or equal to (>=) 9 years on Cycle 1 Day 1 (for all participants) and Cycle 2 and later Day 1 each Cycle (for CNS negative participants); for CNS positive participants: along with MTX, hydrocortisone (HC)/cytarabine (ARA-C) was administered per local standard practice; daratumumab 16 milligrams per kilogram (mg/kg) as intravenous (IV) infusion weekly on Days 1, 8, 15 and 22 of Cycles 1 and 2 then every 2 weeks on Days 1, 15 of Cycle 3 to 6 and every 4 weeks on Day 1 of Cycle 7 and onward; vincristine 1.5 milligrams per meter square (mg/m^2) IV injection/infusion once weekly on Days 1, 8, 15 and 22 of Cycle 1, then every 2 weeks on Days 1 and 15 of Cycle 2 and every 4 weeks on Day 1 of Cycle 3 and onward; prednisone 40 mg/m^2 orally daily on Day 1 to 28 of Cycle 1 and on Day 1 to 5 of Cycle 2 onward. Participants received treatment until disease progression, unacceptable toxicity, or proceeding hematopoietic stem cell transplant after complete response (CR), whichever came first (maximum duration: 2.3 months).
- Cohort 2: T-Cell ALL (1-17 Years): Participants with relapsed/refractory T-cell ALL received intrathecal MTX 8 mg: 1 to <2 years, 10 mg: 2 to <3 years, 12 mg: 3 to <9 years and 15 mg: >=9 years on Cycle 1 Day 1 (all participants) and Cycle 1 Days 15, and 22 (CNS negative participants);for CNS positive participants, along with MTX, HC/ARA-C was administered per local standard practice; daratumumab 16 mg/kg IV infusion weekly on Days 1, 8, 15 and 22 of Cycle 1; doxorubicin 60 mg/m^2 IV infusion once on Day 1; vincristine 1.5 mg/m^2 IV injection/infusion once weekly on Days 1, 8, 15 and 22 on Cycle 1; prednisone 40 mg/m^2 as 2 doses (20 mg/m^2 per dose) orally daily on Day 1 to 28 on Cycle 1; peg-asparaginase 2500 units per meter square (U/m^2) as intramuscular (IM) injection/IV infusion on Days 2, 16 of Cycle 1. In Cycle 2, participants received intrathecal MTX 8 mg: 1 to <2 years, 10 mg: 2 to <3 years, 12 mg: 3 to <9 years and 15 mg: >=9 years on Cycle 2 Days 2 and 15 (CNS negative participants); MTX, HC/ARA-C was administered on Days 2 and 15 per local standard practice (CNS positive participants); daratumumab 16 mg/kg IV infusion weekly on Days 1, 8, 15 and 22; MTX 5 g/m^2 as IV once on Day 2, cyclophosphamide IV 1 g/m^2 once on Day 15; cytarabine 75 mg/m^2 IV/subcutaneous (SC) on Day 16 to 19 and Days 23 to 26; 6-mercaptopurine 60 mg/m^2 orally daily on Days 15 to 28 (maximum duration: 2.9 months).
- Cohort 2: T-Cell ALL (18-30 Years): Participants with relapsed/refractory T-cell ALL in Cycle 1 received intrathecal MTX 8 mg: 1 to <2 years, 10 mg: 2 to <3 years, 12 mg: 3 to <9 years and 15 mg: >=9 years on Cycle 1 Day 1 (all participants) and on Cycle 1 Days 15 and 22 (CNS negative participants); for CNS positive participants, along with MTX, HC/ARA-C was administered per local standard practice; daratumumab 16 mg/kg IV infusion weekly on Days 1, 8, 15 and 22 of Cycle 1; doxorubicin 60 mg/m^2 IV once on Day 1 of Cycle 1; vincristine 1.5 mg/m^2 IV injection/infusion once weekly on Days 1, 8, 15 and 22 of Cycle 1; prednisone 40 mg/m^2 as 2 doses (20 mg/m^2 per dose) orally daily on Days 1 to 28 and peg-asparaginase 2500 U/m^2 as IM injection/IV infusion on Days 2 and 16 of Cycle 1. In Cycle 2, participants received intrathecal MTX 8 mg: 1 to <2 years, 10 mg: 2 to <3 years, 12 mg: 3 to <9 years and 15 mg:>=9 years on Days 2 and 15 (CNS negative participants); MTX, HC/ARA-C was administered on Days 2 and 15 per local standard practice (CNS positive participants); daratumumab 16 mg/kg IV infusion weekly on Days 1, 8, 15 and 22; MTX 5 g/m^2 as IV once on Day 2, cyclophosphamide 1g/m^2 once on Day 15; cytarabine 75 mg/m^2 IV/SC on Days 16 to 19 and Days 23 to 26; and 6-mercaptopurine 60 mg/m^2 orally daily on Days 15 to 28 (maximum duration: 2.1 months).
- Cohort 2: T-Cell Lymphoblastic Leukemia (LL) (1-30 Years): Participants with relapsed/refractory T-cell LL in Cycle 1 received intrathecal MTX 8 mg: 1 to <2 years, 10 mg: 2 to <3 years, 12 mg: 3 to <9 years and 15 mg: >=9 years on Cycle 1 Day 1 (all participants) and on Cycle 1 Days 15 and 22 (CNS negative participants); for CNS positive participants, along with MTX, HC/ARA-C was administered per local standard practice; daratumumab 16 mg/kg IV infusion weekly on Days 1, 8, 15 and 22 of Cycle 1; doxorubicin 60 mg/m^2 IV once on Day 1 of Cycle 1; vincristine 1.5 mg/m^2 IV injection/infusion weekly on Days 1, 8, 15 and 22 of Cycle 1; prednisone 40 mg/m^2 as 2 doses (20 mg/m^2 per dose) orally daily on Days 1 to 28 and peg-asparaginase 2500 U/m^2 as IM injection/IV infusion on Days 2 and 16 of Cycle 1. In Cycle 2, participants received intrathecal MTX 8 mg: 1 to <2 years, 10 mg: 2 to <3 years, 12 mg: 3 to <9 years and 15 mg:>=9 years on Days 2 and 15 (CNS negative participants); MTX, HC/ARA-C was administered by on Days 2 and 15 per local standard practice (CNS positive participants); daratumumab 16 mg/kg IV infusion weekly on Days 1, 8, 15 and 22; MTX 5 g/m^2 as IV once on Day 2, cyclophosphamide 1g/m^2 once on Day 15; cytarabine 75 mg/m^2 IV/SC on Days 16 to 19 and Days 23 to 26; and 6-mercaptopurine 60 mg/m^2 orally daily on Days 15 to 28 (maximum duration: 2.3 months).
Period: Overall Study
Arm/Group | Cohort 1: B-cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (18-30 Years) | Cohort 2: T-Cell Lymphoblastic Leukemia (LL) (1-30 Years)
Started | 7 | 24 | 5 | 10
Completed | 7 | 24 | 4 | 10
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: B-cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (18-30 Years) | Cohort 2: T-Cell Lymphoblastic Leukemia (LL) (1-30 Years) | Total
Number analyzed (Participants) | 7 | 24 | 5 | 10 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.1 (5.01) | 9.8 (4.17) | 22.2 (2.77) | 13.5 (5.68) | 11.7 (6.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 10 | 0 | 1 | 15
  Male | 3 | 14 | 5 | 9 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 2 | 1 | 8
  Not Hispanic or Latino | 4 | 16 | 3 | 7 | 30
  Unknown or Not Reported | 2 | 4 | 0 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 5 | 18 | 2 | 8 | 33
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 0 | 2 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  BELGIUM | 0 | 1 | 0 | 0 | 1
  FRANCE | 0 | 3 | 0 | 2 | 5
  GERMANY | 2 | 0 | 0 | 0 | 2
  ISRAEL | 0 | 2 | 0 | 0 | 2
  ITALY | 2 | 4 | 0 | 0 | 6
  NETHERLANDS | 0 | 2 | 0 | 0 | 2
  SPAIN | 2 | 5 | 1 | 4 | 12
  UNITED KINGDOM | 0 | 3 | 1 | 1 | 5
  UNITED STATES | 1 | 4 | 3 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Percentage of Participants With Complete Response (CR) for B-cell Acute Lymphoblastic Leukemia (ALL)
Description: Complete response based on the modified National Comprehensive Cancer Network (NCCN) criteria was defined as: less than 5 percent (%) blasts in the bone marrow; no evidence of circulating blasts or extramedullary disease; full recovery of peripheral blood counts: platelets greater than (>)100*10^9 cells/liter (L) and absolute neutrophil count (ANC) >1.0*10^9 cells/L. This outcome measure was planned to be analyzed for specified arm only.
Time Frame: Up to 2 cycles, that is, up to 56 days (each cycle of 28-days)
Population: The all treated analysis set included all enrolled participants who received at least 1 dose of daratumumab.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: B-cell ALL (1-17 Years)
Number analyzed (Participants) | 7
Percentage of participants | 0 [NA to NA] — Here, "NA" indicates that lower and upper limit of 90% confidential interval (CI) was not estimable because no participants had the event.

2. Primary Outcome: Cohort 2: Percentage of Participants With Complete Response (CR) for T-cell ALL
Description: Complete response based on the modified NCCN criteria was defined as: less than 5% blasts in the bone marrow; no evidence of circulating blasts or extramedullary disease; full recovery of peripheral blood counts: platelets >100*10^9 cells/L and ANC >1.0*10^9 cells/L. This outcome measure was planned to be analyzed for specified arms only.
Time Frame: End of Cycle 1 (that is, up to 28 days)
Population: The all treated analysis set included all enrolled participants who received at least 1 dose of daratumumab.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2: T-Cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (18-30 Years) | Cohort 2: T-Cell Lymphoblastic Leukemia (LL) (1-30 Years)
Number analyzed (Participants) | 24 | 5 | 10
Percentage of participants | 41.7 [24.6 to 60.3] | 60.0 [18.9 to 92.4] | 30.0 [8.7 to 60.7]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: For ALL participants, ORR was defined as percentage of participants who achieved CR or CR with only partial hematological recovery(CRi) as per NCCN criteria. CR for ALL: less than 5% blasts in bone marrow; no evidence of circulating blasts or extramedullary disease; full recovery of peripheral blood counts: platelets >100*10^9 cells/L and ANC >1.0*10^9 cells/L. CRi for ALL: less than 5% blasts in bone marrow; no evidence of circulating blasts or extramedullary disease; partial recovery of peripheral blood counts not meeting criteria for CR. For LL participants, ORR was defined as percentage of participants who had CR or PR during or after treatment administration but prior to start of subsequent anti-cancer therapy or allogeneic hematopoietic stem cell transplant(HSCT). CR for LL: disappearance of all evidence of disease from all sites. PR for LL: decrease of >=50% in sum of products of diameter of lesions of up to 6 of largest dominant nodes or nodal masses with no new lesions.
Time Frame: Up to 4 years 4 months
Population: The all treated analysis set included all enrolled participants who received at least 1 dose of daratumumab.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: B-cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (18-30 Years) | Cohort 2: T-Cell Lymphoblastic Leukemia (LL) (1-30 Years)
Number analyzed (Participants) | 7 | 24 | 5 | 10
Percentage of participants | 14.3 [0.7 to 52.1] | 83.3 [65.8 to 94.1] | 80.0 [34.3 to 99.0] | 50.0 [22.2 to 77.8]

4. Secondary Outcome: Event-free Survival (EFS)
Description: EFS was defined as the time (in months) from the date of first treatment to the first documented treatment failure (that is [ie], disease progression) or date of relapse from CR or death due to any cause, whichever occurred first. Per NCCN criteria, relapse from CR is defined as: reappearance of leukemia blasts in the peripheral blood or >5% blasts in the bone marrow; reappearance of extramedullary disease or new extramedullary disease. Progressive disease: increase of at least 25% in the absolute number of circulating peripheral or bone marrow blasts, or development of new extramedullary disease. Kaplan-Meier method was used for the analysis.
Time Frame: Up to 4 years 4 months
Population: The all treated analysis set included all enrolled participants who received at least 1 dose of daratumumab.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Cohort 1: B-cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (18-30 Years) | Cohort 2: T-Cell Lymphoblastic Leukemia (LL) (1-30 Years)
Number analyzed (Participants) | 7 | 24 | 5 | 10
Months | 1.1 [0.9 to 2.1] | 8.9 [5.3 to NA] — Here, "NA" indicates that upper limit of 90% CI was not evaluable due to less number of participants with events. | 10.3 [2.6 to NA] — Here, "NA" indicates that upper limit of 90% CI was not evaluable due to less number of participants with events. | 2.9 [1.3 to 4.9]

5. Secondary Outcome: Relapse-free Survival (RFS)
Description: RFS was defined as the time (in months) from CR to relapse from CR, or disease progression or death due to any cause, whichever occurred first. For ALL, as per NCCN criteria, relapse from CR is defined as: reappearance of leukemia blasts in the peripheral blood or >5% blasts in the bone marrow, or reappearance of extramedullary disease or new extramedullary disease. Progressive disease: increase of at least 25% in absolute number of circulating peripheral or bone marrow blasts, or development of new extramedullary disease. Kaplan-Meier method was used for analysis.
Time Frame: Up to 4 years 4 months
Population: The response evaluable analysis set included all enrolled participants who received at least 1 dose of daratumumab and had at least 1 adequate post-baseline disease assessment. Here, 'N' (number of participants analysed) signifies all treated participants who achieved a complete response.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Cohort 1: B-cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (18-30 Years) | Cohort 2: T-Cell Lymphoblastic Leukemia (LL) (1-30 Years)
Number analyzed (Participants) | 0 | 12 | 3 | 4
Months |  | 19.4 [5.3 to NA] — Here, "NA" indicates that upper limit of 90% CI was not evaluable due to less number of participants with events. | 9.4 [3.6 to NA] — Here, "NA" indicates that upper limit of 90% CI was not evaluable due to less number of participants with events. | NA [1.8 to NA] — Here, "NA" indicates that median and upper limit of 90% CI was not evaluable due to less number of participants with events.

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time (in months) from the date of first study drug administration to the date of death due to any cause. Kaplan-Meier method was used for the analysis. Participants who died after consent withdrawal were considered as having an OS event.
Time Frame: Up to 4 years 4 months
Population: The all treated analysis set included all enrolled participants who received at least 1 dose of daratumumab.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Cohort 1: B-cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (18-30 Years) | Cohort 2: T-Cell Lymphoblastic Leukemia (LL) (1-30 Years)
Number analyzed (Participants) | 7 | 24 | 5 | 10
Months | 3.2 [1.0 to 3.6] | 10.9 [6.7 to NA] — Here, "NA" indicates that upper limit of 90% CI was not evaluable due to less number of participants with events. | 12.0 [4.5 to NA] — Here, "NA" indicates that upper limit of 90% CI was not evaluable due to less number of participants with events. | 4.2 [1.7 to 5.6]

7. Secondary Outcome: Minimal Residual Disease (MRD) Negative Rate
Description: MRD negative rate was defined as the percentage of participants who were considered MRD negative after MRD testing by bone marrow aspirate at any timepoint after first study treatment administration and before disease progression or starting subsequent anti-cancer therapy or allogeneic hematopoietic stem cell transplant (HSCT). MRD negative was defined as less than (<) 0.01% abnormal population counts to nucleated mononuclear cells when measured by flow cytometry.
Time Frame: Up to 4 years 4 months
Population: The all treated analysis set included all enrolled participants who received at least 1 dose of daratumumab.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: B-cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (18-30 Years) | Cohort 2: T-Cell Lymphoblastic Leukemia (LL) (1-30 Years)
Number analyzed (Participants) | 7 | 24 | 5 | 10
Percentage of participants | 0 [0 to 0] | 45.8 [28.2 to 64.2] | 20.0 [1.0 to 65.7] | 50.0 [22.2 to 77.8]

8. Secondary Outcome: Percentage of Participants Who Received an Allogeneic Hematopoietic Stem Cell Transplant (HSCT)
Description: Percentage of participants who received an allogeneic HSCT after treatment with daratumumab were reported.
Time Frame: Up to 4 years 4 months
Population: The all treated analysis set included all enrolled participants who received at least 1 dose of daratumumab.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: B-cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (18-30 Years) | Cohort 2: T-Cell Lymphoblastic Leukemia (LL) (1-30 Years)
Number analyzed (Participants) | 7 | 24 | 5 | 10
Percentage of participants | 14.3 [0.7 to 52.1] | 75.0 [56.5 to 88.5] | 60.0 [18.9 to 92.4] | 30.0 [8.7 to 60.7]

9. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Daratumumab
Description: Cmax was defined as maximum observed serum concentration of daratumumab.
Time Frame: Cohort 1: B-cell ALL: End of infusion (EOI) on Day 1 of Cycle 2; Cohort 2: T-cell ALL (1-17 years): EOI on Day 22 of Cycle 2; Cohort 2: T-cell ALL (18-30 years): EOI on Day 1 of Cycle 2; Cohort 2: T-cell LL (1-30 years): EOI on Day 22 of Cycle 2
Population: The serum pharmacokinetics (PK) evaluable analysis set included all enrolled participants who received at least 1 dose of daratumumab and provided at least 1 post-infusion blood sample for serum daratumumab concentrations.
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter (mcg/mL)
Arm/Group | Cohort 1: B-cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (18-30 Years) | Cohort 2: T-Cell Lymphoblastic Leukemia (LL) (1-30 Years)
Number analyzed (Participants) | 7 | 24 | 5 | 10
Micrograms per milliliter (mcg/mL) | 494 (184) | 763 (185) | 501 (347) | 758 (157)

10. Secondary Outcome: Minimum Observed Serum Concentration (Cmin) of Daratumumab
Description: Cmin was defined as minimum observed serum concentration of daratumumab.
Time Frame: Cohort 1: B-cell ALL: Predose on Day 1 of Cycle 2; Cohort 2: T-cell ALL (1-17 years): Predose on Day 22 of Cycle 2; Cohort 2: T-cell ALL (18-30 years): Predose on Day 1 of Cycle 2; Cohort 2: T-cell LL (1-30 years): Predose on Day 22 of Cycle 2
Population: The serum PK evaluable analysis set included all enrolled participants who received at least 1 dose of daratumumab and provided at least 1 post-infusion blood sample for serum daratumumab concentrations.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort 1: B-cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (18-30 Years) | Cohort 2: T-Cell Lymphoblastic Leukemia (LL) (1-30 Years)
Number analyzed (Participants) | 7 | 24 | 5 | 10
mcg/mL | 172 (115) | 369 (105) | 172 (177) | 365 (204)

11. Secondary Outcome: Number of Participants With Anti-daratumumab Antibodies
Description: Number of participants with anti-daratumumab antibodies was reported.
Time Frame: Up to 4 years 4 months
Population: The immunogenicity evaluable analysis set included all enrolled participants who received at least 1 dose of daratumumab and had at least 1 post-infusion sample for detection of anti-daratumumab antibodies.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: B-cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (18-30 Years) | Cohort 2: T-Cell Lymphoblastic Leukemia (LL) (1-30 Years)
Number analyzed (Participants) | 5 | 22 | 5 | 9
Participants | 0 | 0 | 0 | 0

12. Secondary Outcome: Concentration of Daratumumab in Cerebrospinal Fluid (CSF)
Description: Concentration of daratumumab in CSF was reported. '0' in the number analyzed field signifies that none of the participants were available for the analysis at the specified time points.
Time Frame: Pre-dose on Cohort 1: Cycles 1 and 2: Day 1; Cohort 2: Cycle 1 Day 1 and Day 15 and Cycle 2 Day 2 and Day 15
Population: The CSF PK evaluable analysis set included all enrolled participants who received at least 1 dose of daratumumab and provided at least 1 post-infusion CSF sample for daratumumab concentrations. Here, 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure and 'n' (number analyzed) represent number of participants evaluable for specified timepoints.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort 1: B-cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (18-30 Years) | Cohort 2: T-Cell Lymphoblastic Leukemia (LL) (1-30 Years)
Number analyzed (Participants) | 3 | 21 | 5 | 10
mcg/mL
  Cycle 1 Day 1 predose: number analyzed (Participants) | 3 | 18 | 3 | 10
  Cycle 1 Day 1 predose | NA (NA) — Here, "NA" indicates that mean and standard deviation could not calculated due to the lower limit of quantification (LLOQ) limit (0.015 mcg/mL). | NA (NA) — Here, "NA" indicates that mean and standard deviation could not calculated due to the lower limit of quantification (LLOQ) limit (0.015 mcg/mL). | NA (NA) — Here, "NA" indicates that mean and standard deviation could not calculated due to the lower limit of quantification (LLOQ) limit (0.015 mcg/mL). | NA (NA) — Here, "NA" indicates that mean and standard deviation could not calculated due to the lower limit of quantification (LLOQ) limit (0.015 mcg/mL).
  Cycle 1 Day 15 predose: number analyzed (Participants) | 0 | 21 | 5 | 10
  Cycle 1 Day 15 predose |  | 0.907 (1.96) | 0.319 (0.203) | 0.456 (0.280)
  Cycle 2 Day 1 predose: number analyzed (Participants) | 3 | 0 | 0 | 0
  Cycle 2 Day 1 predose | 0.573 (0.545) |  |  |
  Cycle 2 Day 2 predose: number analyzed (Participants) | 0 | 14 | 3 | 5
  Cycle 2 Day 2 predose |  | 0.915 (0.916) | 0.296 (0.191) | 1.23 (0.728)
  Cycle 2 Day 15 predose: number analyzed (Participants) | 0 | 16 | 1 | 5
  Cycle 2 Day 15 predose |  | 0.934 (0.549) | 0.163 | 1.06 (0.282)

ADVERSE EVENTS:
Time Frame: From baseline (Day 1) up to 4 years 4 months
Description: The safety analysis set included all enrolled participants who received at least 1 dose of daratumumab.
Arm/Group | Cohort 1: B-cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (1-17 Years) | Cohort 2: T-Cell ALL (18-30 Years) | Cohort 2: T-Cell Lymphoblastic Leukemia (LL) (1-30 Years)
All-Cause Mortality (participants affected / at risk) | 7/7 | 14/24 | 3/5 | 8/10
Serious Adverse Events (participants affected / at risk) | 3/7 | 16/24 | 4/5 | 7/10
Other Adverse Events (participants affected / at risk) | 7/7 | 24/24 | 5/5 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: B-cell ALL (1-17 Years) (N=7) | Cohort 2: T-Cell ALL (1-17 Years) (N=24) | Cohort 2: T-Cell ALL (18-30 Years) (N=5) | Cohort 2: T-Cell Lymphoblastic Leukemia (LL) (1-30 Years) (N=10)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 | 6 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Anal Fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0
General Physical Health Deterioration (General disorders) | 0 | 1 | 0 | 0
Mucosal Inflammation (General disorders) | 0 | 1 | 0 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 7 | 1 | 1
Hepatic Failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 3 | 0 | 0
Arthritis Bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Campylobacter Infection (Infections and infestations) | 0 | 0 | 0 | 1
Candida Infection (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 0
Enterobacter Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Enterocolitis Infectious (Infections and infestations) | 0 | 1 | 0 | 0
Mucormycosis (Infections and infestations) | 0 | 1 | 0 | 0
Pseudomonas Infection (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0 | 0
Septic Shock (Infections and infestations) | 0 | 2 | 1 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 0
Blood Lactic Acid Increased (Investigations) | 0 | 1 | 0 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 1 | 0 | 0
Pseudomonas Test Positive (Investigations) | 0 | 1 | 0 | 0
Staphylococcus Test Positive (Investigations) | 0 | 1 | 0 | 0
Weight Decreased (Investigations) | 0 | 0 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Brain Oedema (Nervous system disorders) | 0 | 1 | 0 | 0
Depressed Level of Consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0
Leukoencephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral Nerve Palsy (Nervous system disorders) | 0 | 0 | 0 | 1
Posterior Reversible Encephalopathy Syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0
Psychotic Disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 1 | 1
Pharyngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: B-cell ALL (1-17 Years) (N=7) | Cohort 2: T-Cell ALL (1-17 Years) (N=24) | Cohort 2: T-Cell ALL (18-30 Years) (N=5) | Cohort 2: T-Cell Lymphoblastic Leukemia (LL) (1-30 Years) (N=10)
Anaemia (Blood and lymphatic system disorders) | 4 | 16 | 2 | 10
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 7 | 2 | 4
Hypocoagulable State (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 3 | 9 | 1 | 5
Lymph Node Pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 5 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 15 | 2 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 18 | 3 | 9
Cardiac Failure (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 2 | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 2 | 3 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 2
Ear Pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Adrenal Insufficiency (Endocrine disorders) | 0 | 0 | 1 | 1
Eye Oedema (Eye disorders) | 1 | 0 | 0 | 0
Eye Pruritus (Eye disorders) | 0 | 2 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 3 | 0 | 0
Visual Acuity Reduced (Eye disorders) | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 12 | 3 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 3 | 1 | 0
Anal Fissure (Gastrointestinal disorders) | 1 | 3 | 0 | 0
Anal Fistula (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Anal Inflammation (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 6 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 7 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Gingival Bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Lip Dry (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 11 | 2 | 4
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 10 | 2 | 7
Tongue Coated (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 14 | 2 | 5
Asthenia (General disorders) | 0 | 2 | 0 | 0
Catheter Site Haematoma (General disorders) | 0 | 0 | 2 | 0
Chills (General disorders) | 1 | 0 | 1 | 1
Face Oedema (General disorders) | 0 | 2 | 0 | 0
Fatigue (General disorders) | 0 | 3 | 3 | 1
Generalised Oedema (General disorders) | 0 | 3 | 0 | 0
Injection Site Bruising (General disorders) | 0 | 0 | 0 | 1
Localised Oedema (General disorders) | 0 | 1 | 0 | 2
Non-Cardiac Chest Pain (General disorders) | 0 | 2 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 4 | 0 | 3
Pyrexia (General disorders) | 4 | 13 | 3 | 7
Vascular Device Occlusion (General disorders) | 1 | 0 | 0 | 0
Hepatic Cytolysis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 7 | 4 | 4
Drug Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Hypogammaglobulinaemia (Immune system disorders) | 1 | 1 | 0 | 3
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 1
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium Difficile Infection (Infections and infestations) | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1
Device Related Infection (Infections and infestations) | 0 | 2 | 0 | 0
Herpes Simplex (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Kidney Infection (Infections and infestations) | 1 | 0 | 0 | 0
Oral Candidiasis (Infections and infestations) | 0 | 2 | 1 | 1
Otitis Externa (Infections and infestations) | 0 | 2 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1
Periorbital Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Splenic Infection Fungal (Infections and infestations) | 1 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 0 | 0
Vaginal Infection (Infections and infestations) | 0 | 0 | 0 | 1
Accidental Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound Complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 3 | 9 | 3 | 5
Ammonia Increased (Investigations) | 0 | 0 | 1 | 0
Antithrombin Iii Decreased (Investigations) | 0 | 0 | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 2 | 4 | 3 | 5
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 4 | 0
Blood Fibrinogen Decreased (Investigations) | 0 | 3 | 2 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 2 | 0 | 0
Electrocardiogram QT Prolonged (Investigations) | 0 | 0 | 1 | 1
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 3 | 1 | 4
Interleukin Level Increased (Investigations) | 1 | 0 | 0 | 0
International Normalised Ratio Increased (Investigations) | 0 | 0 | 1 | 0
Lipase Increased (Investigations) | 0 | 1 | 2 | 4
Urine Output Decreased (Investigations) | 0 | 0 | 0 | 1
Weight Decreased (Investigations) | 1 | 3 | 2 | 1
Weight Increased (Investigations) | 2 | 0 | 0 | 0
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 4 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Fluid Retention (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperferritinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 5 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 12 | 3 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 8 | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 6 | 4 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 3 | 1 | 2
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 3
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1 | 1
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Depressed Level of Consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 3 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Facial Paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 11 | 2 | 4
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 1 | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 4 | 1 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 2
Device Occlusion (Product Issues) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 2 | 1 | 2
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal Impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal Tubular Disorder (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary Retention (Renal and urinary disorders) | 1 | 1 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Pelvic Pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Allergic Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 0 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 3 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Nasal Mucosal Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Pharyngeal Enanthema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 2
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 4 | 2 | 2
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2
Rash Macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin Striae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 0
Menopause (Social circumstances) | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 2 | 5 | 1 | 4
Hypotension (Vascular disorders) | 0 | 2 | 1 | 2
Superficial Vein Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will with hold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/54/NCT03384654/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/54/NCT03384654/SAP_001.pdf